CLINICAL TRIAL: NCT00976027
Title: Multi-Year Efficacy Study of Fluzone High-Dose Trivalent Vaccine Compared With Fluzone® Vaccine In Adults ≥ 65 Years of Age
Brief Title: Multi-Year Study of Fluzone High-Dose Influenza Vaccine Compared With Fluzone® Vaccine in Adults Aged 65 Years and Older
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No safety concerns, study terminated due to lack of primary endpoint cases in 2009-2010 Flu season (coincided with H1N1 Pandemic) Subjects followed per-protocol
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FIM07; UTN: U1111-1111-4478 (Other: WHO)
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2012-07-25 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Influenza
Keywords: Influenza; Respiratory Tract Infections; Influenza-like illness; Elderly; Fluzone®; Efficacy
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluzone® High Dose Group (Experimental)
  Interventions: Biological: Trivalent inactivated influenza vaccine High Dose
- Fluzone® Group (Active Comparator)
  Interventions: Biological: Trivalent inactivated influenza vaccine

INTERVENTIONS:
Biological: Trivalent inactivated influenza vaccine High Dose — 0.5 mL, Intramuscular
  Other Names: Fluzone® High Dose
  Arms: Fluzone® High Dose Group
Biological: Trivalent inactivated influenza vaccine — 0.5 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Fluzone® Group

SUMMARY:
The aim of this study is to determine the efficacy of Fluzone High Dose vaccine and that of Fluzone® vaccine in the elderly.

Primary objective:

To measure the efficacy of the vaccine, defined as the prevention of laboratory-confirmed influenza caused by viral types/subtypes that are antigenically similar to those contained in the respective annual vaccine formulations.

Secondary objectives:

* To compare the clinical efficacy of Fluzone High Dose vaccine with that of Fluzone® vaccine in elderly adults, with respect to laboratory-confirmed influenza illness caused by any type or subtype of influenza virus.
* To compare the clinical efficacy of Fluzone High Dose vaccine with that of Fluzone® vaccine in elderly adults, in preventing culture-confirmed influenza illness caused by viral types/subtypes antigenically similar to those contained in the respective annual vaccine formulations.

DETAILED DESCRIPTION:
The occurrence of influenza-like illness (ILI) will be determined in elderly participants vaccinated with either Fluzone High Dose or Fluzone® vaccine.

The presence of influenza virus in the respiratory tract of vaccinated individuals with ILI will be confirmed by two methods.

ELIGIBILITY:
Inclusion Criteria :

* Aged ≥ 65 years on the day of vaccination
* Informed consent form signed and dated.
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria :

* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, herbal supplement, or a medical procedure in the 4 weeks preceding the trial vaccination or planned participation in another clinical trial investigating a vaccine, drug, medical device, herbal supplement, or a medical procedure during each year of participation in the study trial.
* Vaccination against influenza in the 6 months preceding the trial vaccination.
* Systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or a history of a life-threatening reaction to Fluzone vaccine or to a vaccine containing any of the same substances.
* Personal history of Guillain-Barré syndrome.
* Dementia or any other cognitive condition at a stage that could interfere with following the trial procedures.
* Thrombocytopenia, bleeding disorder, or anticoagulation therapy contraindicating intramuscular (IM) vaccination.
* Known or suspected human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or Hepatitis C seropositivity.
* Alcohol abuse or drug addiction that could interfere with the subject's ability to comply with trial procedures.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.
* Bedridden subjects.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 9172 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (91):
- United States (89):
  - Birmingham, Alabama
  - Glendale, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tempe, Arizona
  - Fountain Valley, California
  - Los Angeles, California
  - Oceanside, California
  - Sacramento, California
  - Santa Rosa, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Milford, Connecticut
  - Ridgefield, Connecticut
  - Celebration, Florida
  - Clearwater, Florida
  - Coral Gables, Florida
  - Crystal River, Florida
  - Cutler Bay, Florida
  - Deerfield Beach, Florida
  - Inverness, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Sarasota, Florida
  - South Miami, Florida
  - Stockbridge, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - South Bend, Indiana
  - Dubuque, Iowa
  - Arkansas City, Kansas
  - Lenexa, Kansas
  - Lexena, Kansas
  - Newton, Kansas
  - Overland Park, Kansas
  - Prairie Village, Kansas
  - Wichita, Kansas
  - Metairie, Louisiana
  - Columbia, Maryland
  - Elkridge, Maryland
  - Greenbelt, Maryland
  - Brockton, Massachusetts
  - Haverhill, Massachusetts
  - Chaska, Minnesota
  - Edina, Minnesota
  - St Louis, Missouri
  - Missoula, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Rochester, New York
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Akron, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Norman, Oklahoma
  - Corvallis, Oregon
  - Portland, Oregon
  - Downingtown, Pennsylvania
  - Erie, Pennsylvania
  - Jefferson Hills, Pennsylvania
  - Penndel, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Upper Saint Clair, Pennsylvania
  - Anderson, South Carolina
  - Clinton, South Carolina
  - Goose Creek, South Carolina
  - Greer, South Carolina
  - Bristol, Tennessee
  - Nashville, Tennessee
  - Fort Worth, Texas
  - Galveston, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Fredericksburg, Virginia
  - Williamsburg, Virginia
  - Lakewood, Washington
  - Marshfield, Wisconsin
- Puerto Rico (2):
  - San Juan
  - Toa Baja

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study from 22 September 2009 to 07 November 2009 at 99 clinical centers in the US.
Pre-assignment Details: A total of 9158 of the 9172 participants that were randomized were vaccinated, evaluated, and reported in this report.
Groups:
- Fluzone® High Dose: All participants received a single dose of Fluzone High Dose vaccine on Day 0.
- Fluzone®: All subjects received a single dose of Fluzone vaccine on Day 0.
Period: Overall Study
Arm/Group | Fluzone® High Dose | Fluzone®
Started | 6108 | 3050
Completed | 5697 | 2835
Not Completed | 411 | 215
Not completed — Serious Adverse Event | 36 | 17
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 60 | 27
Not completed — Lost to Follow-up | 208 | 103
Not completed — Withdrawal by Subject | 107 | 66

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone® High Dose | Fluzone® | Total
Number analyzed (Participants) | 6108 | 3050 | 9158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 6108 | 3050 | 9158
Age Continuous [Mean (Standard Deviation); unit: Years] | 72.8 (6.0) | 72.8 (5.9) | 72.8 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3268 | 1647 | 4915
  Male | 2840 | 1403 | 4243
Region of Enrollment [Number; unit: Participants]
  United States | 6108 | 3050 | 9158

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Fluzone High Dose Relative to Fluzone in the Prevention of Laboratory Confirmed Influenza Caused by Viral Types and Subtypes That Are Antigenically Similar to Those Contained in the Respective Annual Vaccine Formulations.
Description: The presence (and specific identification) of influenza virus in the respiratory tract of vaccinated individuals with influenza like illness (ILI) was confirmed by tissue culture (for infectious virus) and molecular techniques (polymerase chain reaction based assays), with results reported for cases cause by any viral type or subtype.
Time Frame: Day 0 (pre-vaccination) up to Year 1 post-vaccination
Population: Efficacy was assessed in all participants who met all study inclusion criteria and none of the exclusion criteria, received the vaccine to which they were randomized, and had no protocol violations that might have interfered with evaluation of primary endpoints (Per Protocol Analysis Set).
Measure: Number; unit: Participants
Arm/Group | Fluzone® High Dose | Fluzone®
Number analyzed (Participants) | 6013 | 3008
Participants
  Laboratory Confirmed Cases of ILI | 14 | 8
  Culture Confirmed Cases of ILI | 13 | 7
  PCR Confirmed Cases of ILI | 14 | 8

2. Other Pre Specified Outcome: Number of Participants Reporting Events Associated With All Cases of Protocol Defined Influenza-Like Illness (ILI)
Description: Events associated with Protocol defined influenza-like Illnesses (ILI) were defined as pneumonia, new onset or exacerbation of pre-existing cardio respiratory conditions, health care visits, and medication use (including nonsteroidal anti-inflammatory drugs, NSAIDs).
Time Frame: Day 0 (pre-vaccination) up to the end of the influenza season
Population: The occurrence of events associated with ILI was assessed in all participants who met all study inclusion and exclusion criteria, received the vaccine to which they were randomized, and had no protocol violations that might have interfered with evaluation of primary endpoints (Per-Protocol Analysis Set).
Measure: Number; unit: Participants
Arm/Group | Fluzone® High Dose | Fluzone®
Number analyzed (Participants) | 6013 | 3008
Participants
  Pneumonia | 28 | 14
  Cardio Respiratory Conditions | 10 | 6
  Any Health Care Visit | 478 | 245
  Hospitalization | 31 | 18
  Emergency Room Visit | 40 | 19
  Non Routine Medical Office Visits | 439 | 226
  Any Medication Use (Taken or Prescribed) | 781 | 402
  Antipyretics, NSAIDs, Analgesics Use | 552 | 289
  Antiviral Use | 37 | 12
  Antibiotic Use | 374 | 194

3. Other Pre Specified Outcome: Number of Participants Reporting Events Associated With All Cases of CDC Defined Influenza-Like Illness (ILI)
Description: Events associated with CDC defined influenza-like Illnesses (ILI) were defined as pneumonia, new onset or exacerbation of pre existing cardio respiratory conditions, health care visits, and medication use (including nonsteroidal anti-inflammatory drugs, NSAIDs).
Time Frame: Day 14 (post-vaccination) up to 12 Months post-vaccination
Population: The occurrence of events associated with CDC defined ILI was assessed in all participants who met all study inclusion and exclusion criteria, received the vaccine to which they were randomized, and had no protocol violations that might have interfered with evaluation of primary endpoints (Per-Protocol Analysis Set).
Measure: Number; unit: Participants
Arm/Group | Fluzone® High Dose | Fluzone®
Number analyzed (Participants) | 6013 | 3008
Participants
  Pneumonia | 13 | 7
  New Onset or Exacerbation of Cardio Respiratory | 3 | 1
  Any Health Care Visit | 145 | 82
  Hospitalization | 12 | 6
  Emergency Room Visit | 14 | 9
  Non Routine Medical Office Visits | 129 | 76
  Any Medication Use (Taken or Prescribed) | 220 | 132
  Antipyretics, NSAIDs, Analgesics Use | 153 | 94
  Antiviral Use | 17 | 6
  Antibiotic Use | 123 | 67

4. Other Pre Specified Outcome: Number of Participants Reporting Adverse Events of Special Interest (AESIs) and Serious Adverse Events Post-vaccination With Either Fluzone High-Dose and Fluzone
Description: Adverse events of special interest: new onset of Guillain Barre Syndrome (GBS), Bell's Palsy, encephalitis or myelitis, optic neuritis, Stevens Johnson Syndrome, and toxic epidermal necrolysis
Time Frame: Day 0 before vaccination to Day 180 after vaccination
Population: Adverse events of special interest were assessed in all participants who received study vaccine (Full Analysis Set).
Measure: Number; unit: Participants
Arm/Group | Fluzone® High Dose | Fluzone®
Number analyzed (Participants) | 6108 | 3008
Participants
  Serious Adverse Events (SAE) | 493 | 236
  Death | 31 | 12
  Guillain Barre Syndrome | 0 | 0
  Bell's Palsy | 3 | 2
  Encephalitis or Myelitis | 1 | 0
  Optic Neuritis | 0 | 0
  Stevens Johnson Syndrome | 0 | 0
  Toxic Epidermal Necrolysis | 0 | 0
  SAE Leading to Study Discontinuation | 36 | 17
  Related SAE | 2 | 2
  Related SAE Leading to Study Discontinuation | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 (post-vaccination) up to 8 months post-vaccination.
Arm/Group | Fluzone® High Dose | Fluzone®
Serious Adverse Events (participants affected / at risk) | 493/6108 | 236/3050
Other Adverse Events (participants affected / at risk) | 0/6108 | 0/3050
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluzone® High Dose (N=6108) | Fluzone® (N=3050)
Anaemia (Blood and lymphatic system disorders) | 5 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute Coronary Syndrome (Cardiac disorders) | 0 | 2
Acute Myocardial Infarction (Cardiac disorders) | 3 | 4
Angina Pectoris (Cardiac disorders) | 3 | 5
Angina Unstable (Cardiac disorders) | 7 | 3
Aortic Valve Incompetence (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 16 | 7
Atrioventricular Block Complete (Cardiac disorders) | 2 | 0
Atrioventricular Block First Degree (Cardiac disorders) | 1 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 5 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 3
Cardiac Failure (Cardiac disorders) | 0 | 2
Cardiac Failure Acute (Cardiac disorders) | 1 | 0
Cardiac Failure Chronic (Cardiac disorders) | 1 | 2
Cardiac Failure Congestive (Cardiac disorders) | 20 | 11
Cardiac Valve Disease (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 11 | 4
Coronary Artery Occlusion (Cardiac disorders) | 1 | 0
Coronary Artery Stenosis (Cardiac disorders) | 0 | 1
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 | 1
Mitral Valve Incompetence (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 6 | 8
Myocardial Ischaemia (Cardiac disorders) | 2 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Sick Sinus Syndrome (Cardiac disorders) | 4 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 1
Arteriovenous Malformation (Congenital, familial and genetic disorders) | 0 | 1
Atrial Septal Defect (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 3
Retinal Artery Occlusion (Eye disorders) | 0 | 1
Abdominal Hernia (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 1
Diverticular Perforation (Gastrointestinal disorders) | 3 | 0
Diverticulitis Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 | 0
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer Haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Faeces Discolored (Gastrointestinal disorders) | 0 | 1
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 5 | 3
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus Hernia (Gastrointestinal disorders) | 1 | 0
Ileus Paralytic (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Intestinal Ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 2 | 2
Intestinal Ulcer (Gastrointestinal disorders) | 1 | 0
Intra Abdominal Haematoma (Gastrointestinal disorders) | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Obstruction Gastric (Gastrointestinal disorders) | 0 | 1
Oesophageal Ulcer (Gastrointestinal disorders) | 0 | 1
Oesophageal Ulcer Hemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 7 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 4 | 1
Pancreatitis Relapsing (Gastrointestinal disorders) | 1 | 0
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Reflux Oesophagitis (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 5 | 5
Spigelian Hernia (Gastrointestinal disorders) | 1 | 0
Swollen Tongue (Gastrointestinal disorders) | 1 | 0
Umbilical Hernia Obstructive (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Adverse Drug Reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Catheter Site Haematoma (General disorders) | 1 | 0
Chest Pain (General disorders) | 10 | 9
Chills (General disorders) | 1 | 0
Death (General disorders) | 4 | 0
Fatigue (General disorders) | 0 | 1
Hernia (General disorders) | 1 | 0
Hernia Obstructive (General disorders) | 1 | 0
Influenza Like Illness (General disorders) | 2 | 0
Non Cardiac Chest Pain (General disorders) | 3 | 2
Oedema Peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 4 | 4
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 4 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 2 | 0
Abscess limb (Infections and infestations) | 1 | 0
Actinomycotic pulmonary infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0
Application site cellulitis (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Biliary sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Bronchitis viral (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 9 | 1
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 8 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Sepsis syndrome (Infections and infestations) | 0 | 1
Septic arthritis staphylococcal (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Sialoadenitis (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 8 | 0
Urinary tract infection enterococcal (Infections and infestations) | 2 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 2 | 1
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 4 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 1
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 3 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Medical device complication (Injury, poisoning and procedural complications) | 1 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 3
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 3 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Heart rate irregular (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Back disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 5 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 20 | 9
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hodgkin's disease stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Large cell lung cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Paget's disease of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Splenic neoplasm malignancy unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 4 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 11 | 6
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Drug withdrawal convulsions (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 1
Facial palsy (Nervous system disorders) | 3 | 2
Global amnesia (Nervous system disorders) | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Myelitis transverse (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 2 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 15 | 4
Transient ischaemic attack (Nervous system disorders) | 5 | 5
Alcohol abuse (Psychiatric disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Delusion (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 3 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Incontinence (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 4 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 7 | 3
Renal failure chronic (Renal and urinary disorders) | 1 | 2
Renal mass (Renal and urinary disorders) | 3 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0
Cystocele (Reproductive system and breast disorders) | 2 | 2
Uterine prolapse (Reproductive system and breast disorders) | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 21 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Colectomy (Surgical and medical procedures) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 1 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
Shoulder arthroplasty (Surgical and medical procedures) | 0 | 1
Aneurysm (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 2 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 0
Embolism (Vascular disorders) | 1 | 0
Femoral artery embolism (Vascular disorders) | 0 | 1
Femoral artery occlusion (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 2 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 1
Ischaemia (Vascular disorders) | 0 | 1
Ischaemic limb pain (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 2 | 0
Vascular rupture (Vascular disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 4 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 2 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 3 | 1
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 16 | 13
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to lack of primary endpoint cases in 2009-2010 influenza season (coincided with the H1N1 Pandemic). There were no safety concerns; enrolled subjects were followed per-protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications